CLINICAL TRIAL: NCT03473847
Title: Repeatability and Reproducibility of Carl Zeiss Meditec Cirrus HD OCT 5000, Optovue RTVue OCT, CSO MS-39 OCT and ArcScan Insight 100 Very High-frequency Digital Ultrasound and Comparison Between Devices
Brief Title: Repeatability, Reproducibility and Comparison of Cirrus OCT, RTVue OCT, MS-39 OCT, and Insight 100 VHFDU
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices currently awaiting software updates
Sponsor: London Vision Clinic (Other)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LOVC-006
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Corneal Thickness Measurement; Epithelial Thickness Measurement; LASIK Flap Thickness Measurement; SMILE Cap Thickness Measurement
Keywords: VHF digital ultrasound; Optical coherence tomography; Corneal thickness; Epithelial thickness; LASIK; SMILE

STUDY DESIGN:
Intervention Model Description: Scans from 4 devices obtained on the same patient population for comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Repeatability and Reproducibility - Normal eyes (Experimental): This arm will include 20 eyes of 20 patients with no previous ocular surgery.
  The research participant will be scanned a number of times using each of the four devices (the Insight 100 VHF digital ultrasound scanner, the Cirrus HD OCT 5000, the RTVue OCT, and the MS-39 OCT). The scan sequence will be undertaken on a single day as follows:
  1. 5 consecutive repeated scans of the cornea will be performed by the first operator using each of the four devices (expected total time approximately 5 minutes for each OCT scan set and 15 minutes for the Insight 100 scan set).
  2. There will be a break of about 30 minutes.
  3. 5 consecutive repeated scans of the cornea will be performed by the second operator using each of the four devices (expected total time approximately 5 minutes for each OCT scan set and 15 minutes for the Insight 100 scan set).
  Interventions: Device: ArcScan Insight 100 very high-frequency digital ultrasound; Device: Carl Zeiss Meditec Cirrus HD OCT 5000; Device: Optovue RTVue OCT; Device: CSO MS-39 OCT
- Repeatability and Reproducibility - Post-op eyes (Experimental): This arm will include 20 eyes of 20 patients between 3 and 9 months after corneal laser refractive surgery.
  The research participant will be scanned a number of times using each of the four devices (the Insight 100 VHF digital ultrasound scanner, the Cirrus HD OCT 5000, the RTVue OCT, and the MS-39 OCT). The scan sequence will be undertaken on a single day as follows:
  1. 5 consecutive repeated scans of the cornea will be performed by the first operator using each of the four devices (expected total time approximately 5 minutes for each OCT scan set and 15 minutes for the Insight 100 scan set).
  2. There will be a break of about 30 minutes.
  3. 5 consecutive repeated scans of the cornea will be performed by the second operator using each of the four devices (expected total time approximately 5 minutes for each OCT scan set and 15 minutes for the Insight 100 scan set).
  Interventions: Device: ArcScan Insight 100 very high-frequency digital ultrasound; Device: Carl Zeiss Meditec Cirrus HD OCT 5000; Device: Optovue RTVue OCT; Device: CSO MS-39 OCT
- Comparison between devices - Normal eyes (Experimental): This arm will include 101 eyes of 101 patients with no previous ocular surgery.
  The research participant will be scanned once using each of the four devices (the Insight 100 VHF digital ultrasound scanner, the Cirrus HD OCT 5000, the RTVue OCT, and the MS-39 OCT). Expected total time approximately 20 minutes to complete all four scans.
  Interventions: Device: ArcScan Insight 100 very high-frequency digital ultrasound; Device: Carl Zeiss Meditec Cirrus HD OCT 5000; Device: Optovue RTVue OCT; Device: CSO MS-39 OCT
- Comparison between devices - Post-op eyes (Experimental): This arm will include 101 eyes of 101 patients between 3 and 9 months after corneal laser refractive surgery.
  The research participant will be scanned once using each of the four devices (the Insight 100 VHF digital ultrasound scanner, the Cirrus HD OCT 5000, the RTVue OCT, and the MS-39 OCT). Expected total time approximately 20 minutes to complete all four scans.
  Interventions: Device: ArcScan Insight 100 very high-frequency digital ultrasound; Device: Carl Zeiss Meditec Cirrus HD OCT 5000; Device: Optovue RTVue OCT; Device: CSO MS-39 OCT

INTERVENTIONS:
Device: ArcScan Insight 100 very high-frequency digital ultrasound — The ArcScan Insight 100 VHF digital ultrasound scanner can measure individual layers within the cornea with very high precision, as well as being able to image the interior of the eye including the chamber between the iris and the cornea, the lens and other structures behind the iris. The ArcScan Insight 100 device is a digital ultrasound scanner, meaning that it uses ultrasound waves to measure parameters of the eye. The Insight examination involves the patient sitting in front of the ultrasound unit and looking through a disposable goggle-like eyepiece at a light source. Warm sterile balanced saline solution (like natural tears) are used to fill the space between the light source and the eye, to allow ultrasound transmission. There is no contact between the instrument and the eye other than being immersed in this water bath.
  Other Names: Artemis very high-frequency digital ultrasound
Device: Carl Zeiss Meditec Cirrus HD OCT 5000 — The Cirrus HD OCT 5000 uses high definition spectral domain optical coherence tomography (OCT) to measure anatomical structures of the eye. OCT is non-contact and uses light, rather than ultrasound, to obtain cross-sectional images. An OCT scan involves the patient sitting in front of the device, placing their chin on a chin-rest and fixating on a light source. Nothing comes into contact with the eye and the patient is only aware of the instrument rotating in front of them.
Device: Optovue RTVue OCT — The Optovue RTVue OCT uses high definition Fourier/spectral domain optical coherence tomography (OCT) to measure anatomical structures of the eye. OCT is non-contact and uses light, rather than ultrasound, to obtain cross-sectional images. An OCT scan involves the patient sitting in front of the device, placing their chin on a chin-rest and fixating on a light source. Nothing comes into contact with the eye and the patient is only aware of the instrument rotating in front of them.
Device: CSO MS-39 OCT — The CSO MS-39 OCT uses high definition Fourier domain optical coherence tomography (OCT) to measure anatomical structures of the eye. OCT is non-contact and uses light, rather than ultrasound, to obtain cross-sectional images. The MS-39 also includes a Placido topographer within the device to simultaneously obtain a measurement of the shape (curvature) of the front surface of the cornea, which is then combined with the OCT thickness measurement to generate the shape of the back surface of the cornea.
  An OCT scan involves the patient sitting in front of the device, placing their chin on a chin-rest and fixating on a light source. Nothing comes into contact with the eye and the patient is only aware of the instrument rotating in front of them.

SUMMARY:
The purpose of this study is to evaluate the repeatability and reproducibility of corneal, epithelial, and LASIK flap thickness using the Carl Zeiss Meditec Cirrus HD OCT 5000, Optovue RTVue OCT, CSO MS-39 OCT, and ArcScan Insight 100 very high-frequency digital ultrasound arc-scanner.

DETAILED DESCRIPTION:
Very high-frequency (VHF) digital ultrasound was first used in 1993 to obtain images and measure the thickness of the cornea (the window at the front of the eye) and the layers within the cornea, such as the epithelium (the layer of skin on the surface of the cornea). A commercially available instrument, known as the Artemis, has been used in routine clinical practice since 2001. The ArcScan Insight 100 VHF digital ultrasound scanner is an updated version, which obtained CE mark in 2016.

Optical coherence tomography (OCT) is another method of measuring the thickness of the cornea and the corneal epithelium. OCT has been used for measuring corneal thickness since 1997 and the technology had evolved to also measure epithelial thickness since 2012. There are currently three OCT scanners capable of measuring epithelial thickness; Carl Zeiss Meditec Cirrus HD OCT 5000, Optovue RTVue OCT, CSO MS-39 OCT.

The aim of the study is to establish the repeatability (i.e. the variability in measurements taken by a single examiner during a single visit) and reproducibility (i.e. the variability in measurements taken in the same conditions between two examiners) for each of the four devices for measuring corneal thickness and epithelial thickness.

ELIGIBILITY:
Inclusion Criteria:

Only patients who are medically suitable for corneal laser refractive surgery can be included in the study.

As general inclusion criteria the following aspects are defined:

* Subjects should be 21 years of age or older.
* Contact lens wearers must stop wearing their contact lenses at least four weeks per decade of wear before baseline measurements in case of hard contact lenses and one week before baseline measurements in case of soft contact lenses.
* Patient will be able to understand the patient information and willing to sign an informed consent.

For the normal eye populations:

* Eyes with no ocular pathology
* Eyes with no previous ocular or corneal surgery

For the post-op eye populations:

• Eyes between 3 and 9 months after LASIK or SMILE

Exclusion Criteria:

* Previous ocular or corneal surgery (for normal eyes)
* Patient not being able to tolerate local or topical anesthesia
* Patient has active conjunctivitis or any active ocular infection or inflammation
* Patient has a corneal ulcer
* Patient has an open wound on the corneal epithelium
* Patient has compromised epithelium (e.g. ≥Grade 3 superficial punctate keratitis)
* Pregnancy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Repeatability and reproducibility of Cirrus HD OCT 5000 corneal scans in normal eyes (standard deviation) | 10 minutes (5 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in normal eyes with no previous corneal surgery
Repeatability and reproducibility of RTVue OCT corneal scans in normal eyes (standard deviation) | 10 minutes (5 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in normal eyes with no previous corneal surgery
Repeatability and reproducibility of MS-39 OCT corneal scans in normal eyes (standard deviation) | 10 minutes (5 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in normal eyes with no previous corneal surgery
Repeatability and reproducibility of Insight 100 VHF digital ultrasound corneal scans in normal eyes (standard deviation) | 30 minutes (15 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in normal eyes with no previous corneal surgery
Repeatability and reproducibility of Cirrus HD OCT 5000 corneal scans in post-op eyes (standard deviation) | 10 minutes (5 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in eyes between 3 and 9 months after corneal laser refractive surgery
Repeatability and reproducibility of RTVue OCT corneal scans in post-op eyes (standard deviation) | 10 minutes (5 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in eyes between 3 and 9 months after corneal laser refractive surgery
Repeatability and reproducibility of MS-39 OCT corneal scans in post-op eyes (standard deviation) | 10 minutes (5 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in eyes between 3 and 9 months after corneal laser refractive surgery
Repeatability and reproducibility of Insight 100 VHF digital ultrasound corneal scans in post-op eyes (standard deviation) | 30 minutes (15 minutes per observer)
  The within-observer standard deviation (repeatability) and between-observer standard deviation (reproducibility) calculated by ANOVA for 5 repeated measurements by two observers of corneal thickness and epithelial thickness in eyes between 3 and 9 months after corneal laser refractive surgery
Difference in corneal thickness measurements between Cirrus HD OCT 5000, RTVue OCT, MS-39 OCT, and Insight 100 VHF digital ultrasound in normal eyes | 20 minutes for all four scans
  The difference between each pair of devices for measurements of corneal thickness and epithelial thickness in eyes with no previous ocular surgery.
Difference in corneal thickness measurements between Cirrus HD OCT 5000, RTVue OCT, MS-39 OCT, and Insight 100 VHF digital ultrasound in post-op eyes | 20 minutes for all four scans
  The difference between each pair of devices for corneal thickness, epithelial thickness and interface thickness in eyes between 3 and 9 months after corneal laser refractive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dan Z Reinstein, MD, MA, FRCOphth, Principal Investigator — London Vision Clinic
Locations (1):
- London Vision Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Background] Reinstein DZ, Archer TJ, Gobbe M, Silverman RH, Coleman DJ. Repeatability of layered corneal pachymetry with the artemis very high-frequency digital ultrasound arc-scanner. J Refract Surg. 2010 Sep;26(9):646-59. doi: 10.3928/1081597X-20091105-01. Epub 2009 Nov 16. PMID 19928698
- [Background] Reinstein DZ, Yap TE, Archer TJ, Gobbe M, Silverman RH. Comparison of Corneal Epithelial Thickness Measurement Between Fourier-Domain OCT and Very High-Frequency Digital Ultrasound. J Refract Surg. 2015 Jul;31(7):438-45. doi: 10.3928/1081597X-20150623-01. PMID 26186562
- [Background] Yap TE, Archer TJ, Gobbe M, Reinstein DZ. Comparison of Central Corneal Thickness Between Fourier-Domain OCT, Very High-Frequency Digital Ultrasound, and Scheimpflug Imaging Systems. J Refract Surg. 2016 Feb;32(2):110-6. doi: 10.3928/1081597X-20151223-01. PMID 26856428
- [Background] Kiraly L, Stange J, Kunert KS, Sel S. Repeatability and Agreement of Central Corneal Thickness and Keratometry Measurements between Four Different Devices. J Ophthalmol. 2017;2017:6181405. doi: 10.1155/2017/6181405. Epub 2017 Mar 5. PMID 28357136